CLINICAL TRIAL: NCT01725750
Title: Treatment of Post-TBI Fatigue With Light Therapy
Brief Title: Treatment of Post-Traumatic Brain Injury (Post-TBI) Fatigue With Light Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Kristen Dams-O'Connor, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 12-1256; HSM 12-00759; H133A120084 (Other Grant/Funding Number: National Institute on Disability and Rehabilitation Research)
Record Dates: First submitted 2012-11-07; First posted 2012-11-14 (Estimated); Results first posted 2018-09-11 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-07

CONDITIONS: Traumatic Brain Injury; Fatigue
Keywords: Traumatic Brain Injury; TBI; Fatigue; Post-TBI Fatigue; PTBIF; Depressed Mood; Excessive Daytime Sleepiness; Circadian Rhythm; Anxiety; Cognitive Dysfunction; Intervention; Treatment
MeSH Terms: conditions — Brain Injuries, Traumatic; Fatigue; Consciousness Disorders; Disorders of Excessive Somnolence; Anxiety Disorders; Cognitive Dysfunction | interventions — Ultraviolet Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Bright White Light (BWL) (Experimental): Participants will self-administer bright white light daily using a Litebook® (The Litebook Company Ltd.). The Litebook is a small (6" x 5" x 1") and lightweight (8 oz.) box.
  Interventions: Device: Bright White Light (BWL)
- Dim Red Light (DRL) (Active Comparator): Participants will self-administer dim red light daily using a device that appears identical to Bright White Light (BWL) Litebook but that uses red LEDs emitting DRL.
  Interventions: Device: Dim Red Light (DRL)

INTERVENTIONS:
Device: Bright White Light (BWL) — Participants will self-administer bright white light daily. Litebooks used for Bright White Light and Dim Red Light are identical except for the light which they emit. Users are instructed to place it about 18" from their face and within 45º of the visual field for 30 minutes within half an hour of waking each morning, for 4 weeks. The participant may eat, read, watch TV, etc. while sitting in front of the box.
  Other Names: Litebook - Bright White Light
  Arms: Bright White Light (BWL)
Device: Dim Red Light (DRL) — A device that appears identical to BWL Litebook but that uses red LEDs emitting DRL. Users are instructed to place it about 18" from their face and within 45º of the visual field for 30 minutes within half an hour of waking each morning, for 4 weeks. The participant may eat, read, watch TV, etc. while sitting in front of the box.
  Other Names: Litebook - Dim Red Light
  Arms: Dim Red Light (DRL)

SUMMARY:
This study aims to evaluate the efficacy of 4 weeks of daily light exposure in reducing Post-Traumatic Brain Injury (TBI) Fatigue immediately post-treatment and at a one-month follow up. The investigators hypothesize that individuals receiving 4 weeks of bright white light treatment will report significant reductions in fatigue compared to individuals receiving dim red light treatment for the same duration of time, and that these treatment effects will be maintained one month after treatment completion.

DETAILED DESCRIPTION:
To determine the efficacy of bright white light exposure compared to dim red light exposure in reducing post-TBI fatigue, an 8-week, randomized parallel-group clinical trial will be performed. Outcome assessment will be blinded. Participants will complete a baseline battery (T1) including 72 hours of actigraphy. Participants will then be randomized to either the Bright White Light (BWL) or the Dim Red Light (DRL) group. After 4 weeks of daily, 30-minute light treatments, the baseline battery will be re-administered (T2) along with 3 more days of Actigraphy. A follow-up assessment involving the same measures will be administered 1 month-post cessation of light therapy (T3). Participant treatment allocations will be masked for research team members conducting outcome measures. Secondary outcome measures will be administered to explore the effects of light therapy on mood, daytime sleepiness, sleep quality, circadian rhythms, anxiety, cognition and life satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Documented TBI of any severity
* At least 6 months post injury
* Presence of clinically significant fatigue, operationalized as a score of 22 or more on the Multidimensional Assessment of Fatigue
* Age 18 or older
* English speaking

Exclusion Criteria:

* Neurological disease other than TBI
* Pregnancy (because of pregnancy fatigue)
* Medical illness causing fatigue, such as anemia, hypothyroidism, HIV, renal failure, cirrhosis or cancer treatment in the past year
* Current major depressive episode or substance abuse
* Diagnosed sleep disorder or high risk for sleep apnea
* History of bipolar disorder or manic or hypomanic episodes
* Current chronic, severe headaches
* Sensitivity to bright light
* History of retinal damage or disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Gordon, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Kirsten Dams-O'Connor, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- The Brain Injury Research Center at Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From October 2015-January 2017, recruitment materials were sent to previous research and support group participants, and other local TBI centers. Information was also posted online and at consumer conferences. External sites included Centre for Neuro Skills facilities and post-acute rehab centers in Bakersfield and Los Angeles, CA, and Dallas, TX.
Period: Overall Study
Arm/Group | Bright White Light (BWL) | Dim Red Light (DRL)
Started | 44 | 44
Completed | 42 | 34
Not Completed | 2 | 10
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 0 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bright White Light (BWL) | Dim Red Light (DRL) | Total
Number analyzed (Participants) | 44 | 44 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.045 (16.335) | 45.182 (13.138) | 46.614 (14.808)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 44
  Male | 24 | 20 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian/Pacific Islander | 2 | 5 | 7
  Hispanic/Latino | 5 | 8 | 13
  Black or African American | 6 | 5 | 11
  White | 27 | 23 | 50
  More than one race/Other | 4 | 3 | 7
Years of education completed [Mean (Standard Deviation); unit: years] | 15.841 (2.533) | 15.651 (2.654) | 15.747 (2.580)

OUTCOME MEASURES:

1. Primary Outcome: Multidimensional Assessment of Fatigue (MAF)
Description: Multidimensional Assessment of Fatigue (MAF) yields a Global Fatigue Index (GFI), assessing 5 dimensions of fatigue: distress, degree, severity, impact on ADLs and frequency of fatigue in the past week, and it yields a composite score. GFI full score from 0-50, with a higher score indicating more severe fatigue, fatigue distress, or impact on activities of daily living.
Time Frame: baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bright White Light (BWL) | Dim Red Light (DRL)
Number analyzed (Participants) | 44 | 44
score on a scale
  Baseline | 33.332 (9.043) | 30.531 (10.633)
  4 weeks (end of treatment) | 27.993 (9.993) | 24.937 (10.558)
  8 weeks (one month post treatment) | 28.658 (12.213) | 25.350 (10.895)

2. Secondary Outcome: TBI-QOL Fatigue
Description: The Traumatic Brain Injury-Quality Of Life Fatigue (TBI-QOL) measures form part of the Promis Neuro-QOL initiative and include well-validated self-report measures that assess the health-related QOL of individuals with neurological disorders. All TBI-QOL scores have been transformed to a T metric,from 0-100, with a mean of 50 (SD = 10), with a higher score indicating more fatigue.
Time Frame: baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Bright White Light (BWL) | Dim Red Light (DRL)
Number analyzed (Participants) | 44 | 44
T score
  Baseline | 61.819 (6.255) | 58.821 (7.533)
  4 weeks (end of treatment) | 58.071 (7.384) | 55.724 (8.305)
  8 weeks (one month post treatment) | 58.226 (8.481) | 57.252 (9.033)

3. Secondary Outcome: Neuro-QOL Depression and Sleep
Description: The Neuro-QOL Depression and Sleep measures the physical, mental, and social effects experienced by adults and children living with neurological conditions. Raw scores were converted to T-Scores; from 0-100, with a T = 50 indicating average function compared to the reference population and a standard deviation of 10, with a higher score indicating worse function.
Time Frame: baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Bright White Light (BWL) | Dim Red Light (DRL)
Number analyzed (Participants) | 44 | 44
T-score
  Baseline | 52.893 (8.033) | 82.942 (7.570)
  4 weeks (end of treatment) | 53.337 (8.190) | 52.864 (7.896)
  8 weeks (one month post treatment) | 55.162 (8.193) | 52.290 (9.698)

4. Secondary Outcome: Epworth Sleepiness Scale (ESS)
Description: The Epworth Sleepiness Scale (ESS) will also be used, to assess daytime sleepiness; it is an 8-item measure that asks about the probability of dozing or sleeping during typical daytime activities and has been widely used in TBI research. Scores correlate well with objective measures of speed of daytime sleep onset. The test is a list of eight situations in which the participate rates tendency to become sleepy on a scale of 0, no chance of dozing, to 3, high chance of dozing for each item. Total scale from 0 to 24, with higher score indicating severe excessive daytime sleepiness.
Time Frame: baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bright White Light (BWL) | Dim Red Light (DRL)
Number analyzed (Participants) | 44 | 44
score on a scale
  baseline | 9.695 (4.869) | 6.970 (4.323)
  4 weeks (end of treatment) | 8.162 (3.927) | 8.312 (3.182)
  8 weeks (one month post treatment) | 8.169 (4.041) | 8.133 (3.899)

5. Secondary Outcome: CNS Vital Signs TBI Rehab Toolbox
Description: The Centre for Neuro Skills Vital Signs TBI Rehab Toolbox is a brief, 25-minute computerized cognition battery; it emphasizes those cognitive functions that are the most likely to respond to alerting effects of light (vigilance, attention, speed) and has multiple forms for serial assessment. The scores are reported as Standard Scores, with mean = 100 and standard deviation = 15. Higher scores are correlated with better outcomes.
Time Frame: baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bright White Light (BWL) | Dim Red Light (DRL)
Number analyzed (Participants) | 44 | 44
score on a scale
  baseline | 79.59 (26.260) | 82.83 (21.805)
  4 weeks (end of treatment) | 83.19 (27.489) | 77.64 (37.658)
  8 weeks (one month post treatment) | 86.17 (28.051) | 79.10 (35.443)

6. Secondary Outcome: Cognitive Failures Questionnaire
Description: The Cognitive Failures Questionnaire (CFQ)100 is a 25-item self-report inventory, with items measuring difficulties in several cognitive domains (e.g., memory, perception), each item scored from 0 (never) to 4 (very often), with total scale from 0 - 100, with higher score indicating worse outcome.
Time Frame: baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bright White Light (BWL) | Dim Red Light (DRL)
Number analyzed (Participants) | 44 | 44
score on a scale
  baseline | 47.823 (16.872) | 42.806 (15.175)
  4 weeks (end of treatment) | 45.261 (17.590) | 46.564 (16.646)
  8 weeks (one month post treatment) | 47.503 (18.204) | 45.352 (18.310)

7. Secondary Outcome: Neuro-QOL Anxiety
Description: The Neuro-QOL Anxiety measure. Raw scores were converted to T-Scores; from 0-100, with a T = 50 indicating average function compared to the reference population and a standard deviation of 10, with a higher score indicating worse anxiety.
Time Frame: baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Bright White Light (BWL) | Dim Red Light (DRL)
Number analyzed (Participants) | 44 | 44
T score
  baseline | 55.725 (8.137) | 56.253 (7.581)
  4 weeks (end of treatment) | 55.250 (8.929) | 56.661 (7.766)
  8 weeks (one month post treatment) | 57.441 (8.073) | 55.226 (8.828)

8. Secondary Outcome: Actiwatch Spectrum - Acrophase
Description: Philips Actiwatch Spectrum to measure circadian rhythms; it is the size and shape of a digital wristwatch and weighs about one ounce. It is worn on an ordinary watchband and is waterproof. Data can be downloaded and analyzed using Actiware software. The Actiwatch Spectrum logs all physical movement using a piezoelectric accelerometer and detects the presence of ambient light (400-700nm), making it a useful measure of circadian cycles because it allows for accurate quantitative assessment of periods of activity, rest and sleep.
  Acrophase is time of the peak activity, so it is expressed in hours. The higher the number, the later in the day the peak activity occurs.
Time Frame: 4 weeks post treatment
Population: After the Actigraph data were cleaned and analyzed, there was clean, usable data for 30 in the white arm and 23 in the red arm.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Bright White Light (BWL) | Dim Red Light (DRL)
Number analyzed (Participants) | 30 | 23
hours | 15.68 (2.29) | 15.98 (1.09)

9. Secondary Outcome: Actiwatch Spectrum - Mesor
Description: Philips Actiwatch Spectrum to measure circadian rhythms; it is the size and shape of a digital wristwatch and weighs about one ounce. It is worn on an ordinary watchband and is waterproof. Data can be downloaded and analyzed using Actiware software. The Actiwatch Spectrum logs all physical movement using a piezoelectric accelerometer and detects the presence of ambient light (400-700nm), making it a useful measure of circadian cycles because it allows for accurate quantitative assessment of periods of activity, rest and sleep.
  Mesor is an adjusted proportion of the difference between the minimum and half the peak, so range is 0-1. Higher means a more rhythmic pattern.
Time Frame: 4 weeks post treatment
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bright White Light (BWL) | Dim Red Light (DRL)
Number analyzed (Participants) | 30 | 23
score on a scale | 0.72 (0.21) | 0.83 (0.25)

10. Secondary Outcome: Actiwatch Spectrum - F Statistic
Description: Philips Actiwatch Spectrum to measure circadian rhythms; it is the size and shape of a digital wristwatch and weighs about one ounce. It is worn on an ordinary watchband and is waterproof. Data can be downloaded and analyzed using Actiware software. The Actiwatch Spectrum logs all physical movement using a piezoelectric accelerometer and detects the presence of ambient light (400-700nm), making it a useful measure of circadian cycles because it allows for accurate quantitative assessment of periods of activity, rest and sleep.
  F statistic is an F value, so the range is 0 - infinity. It compares two different models of calculating the curve. Higher means a more rhythmic pattern.
Time Frame: 4 weeks post treatment
Population: After the Actigraph data were cleaned and analyzed, there was clean, usable data for 30 in the white arm and in the 23 red arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bright White Light (BWL) | Dim Red Light (DRL)
Number analyzed (Participants) | 30 | 23
score on a scale | 1765.36 (1120.32) | 2307.38 (1574.54)

11. Secondary Outcome: Satisfaction With Life Scale
Description: Satisfaction with Life Scale, a 5-item measure of global satisfaction with life, on likert scale from 1 strongly disagree to 7 strongly agree. Total scale from 5 to 35, with higher scores indicating more satisfaction with life, and 20 representing a neutral point on the scale.
Time Frame: baseline, 4 weeks, 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bright White Light (BWL) | Dim Red Light (DRL)
Number analyzed (Participants) | 44 | 44
score on a scale
  baseline | 17.409 (6.956) | 18.698 (7.386)
  4 weeks (end of treatment) | 17.622 (7.154) | 18.394 (7.925)
  8 weeks (one month post treatment) | 17.441 (6.219) | 19.900 (6.707)

12. Secondary Outcome: Treatment Satisfaction Questionnaire for Medication
Description: An adapted version of the Treatment Satisfaction Questionnaire for Medication (TSQM). This is a validated, psychometrically sound measure of general treatment satisfaction. The TSQM scores range from 0 to 100 with higher scores representing higher satisfaction.
Time Frame: at 4 weeks (end-of-treatment)
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Bright White Light (BWL) | Dim Red Light (DRL)
Number analyzed (Participants) | 44 | 44
score on a scale | 42.455 (29.827) | 47.546 (33.112)

13. Secondary Outcome: Credibility/Expectancy Questionnaire
Description: Assess treatment credibility (BWL vs. DRL) with the Credibility/Expectancy Questionnaire (CEQ), used in clinical outcome studies. The CEQ utilizes two scales during the administration (1-9, and 0-100%), and so a composite z score was derived for each factor (expectancy and credibility) by first standardizing the individual items and then summing those items for each factor. The Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean. A higher score indicates more belief or feeling of reduction in anxiety.
Time Frame: at 4 weeks (end-of-treatment)
Population: Compared to other outcome measures, fewer CEQ records were analyzed due to participant non-compliance.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bright White Light (BWL) | Dim Red Light (DRL)
Number analyzed (Participants) | 43 | 37
score on a scale | -.5539 (2.577) | .4489 (2.74)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Bright White Light (BWL) | Dim Red Light (DRL)
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/44
Other Adverse Events (participants affected / at risk) | 1/44 | 0/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bright White Light (BWL) (N=44) | Dim Red Light (DRL) (N=44)
Blurred vision (Eye disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT01725750/Prot_SAP_000.pdf